CLINICAL TRIAL: NCT06006988
Title: Investigation of the Relationship Between Trunk Control and Viscoelastic Properties of Trunk Muscles in Acute Stroke Patients
Brief Title: Trunk Control and Viscoelastic Properties of Trunk Muscles in Acute Stroke Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sanko University (Other)
Responsible Party: Principal Investigator, Hakan Polat, Director, Sanko University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: DrHakanPolat
Record Dates: First submitted 2023-08-01; First posted 2023-08-23 (Actual); Last update posted 2023-08-23 (Actual); Status verified 2023-08

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- trunk disorder scale (Experimental): It is a 17-parameter scale developed for the evaluation of trunk control. Existing sections in the scale; static sitting balance (GBÖ Static), dynamic sitting balance (GBÖ Dynamic) and coordination (GBÖ Coordination). The total score is a minimum of 0 and a maximum of 23 points and it is accepted that the higher score shows better performance.
  Interventions: Combination Product: myoton pro

INTERVENTIONS:
Combination Product: myoton pro — MyotonPRO is a mobile, removable handheld myotonometer. This tool is noninvasive and provides a quantitative assessment of a muscle's viscoelastic properties. These properties are characterized by various parameters such as hardness, tone and elasticity. The probe of MyotonPRO delivers a short (15 ms), low intensity (0.58 N) mechanical impact/impact on the skin on the muscle. The response of the touch then generates a recorded signal and an internal software program generates an acceleration graph. Measurements of various viscoelastic muscle properties such as stiffness, tone and elasticity are then extracted from this graph.

SUMMARY:
Stroke is a health problem that ranks second among the causes of death and third in the rate of severe disability . One of the most commonly reported problems after stroke is the structural and functional changes in the muscles . At the beginning of the structural changes of the muscles is the effect of the viscoelastic properties of the muscles. Various studies have reported an increase in skeletal muscle stiffness, which is dependent on elasticity as well as muscle viscosity after stroke . The initial condition of the affected trunk on both the ipsilateral and contralateral sides after stroke is defined as the earliest and most important factor in predicting functional recovery. Functional recovery after stroke was found to be associated with trunk control at a rate of 45-71% in general . We think that viscoelastic properties will change in trunk muscles of individuals with acute stroke and these changes may be related to trunk control disorder.

DETAILED DESCRIPTION:
Trunk control is the ability to maintain an upright posture, adjust weight shift, and perform selective movements in the trunk to keep the center of gravity within the base of support . Stroke is one of the main causes of impaired trunk control, including center of gravity and balance reaction . In stroke patients, trunk control ability is decreased in all planes, especially in the frontal plane. Studies have reported that stroke patients have a decrease in trunk muscle strength compared to healthy individuals , and when trunk proprioception is measured in chronic stroke patients, it is affected more than healthy participants . In addition, skeletal muscles undergo various changes after stroke. These changes that occur in the musculoskeletal system are muscle weakness, fatigue, and abnormal muscle tone . Changes at the muscle level include tissue elasticity and viscous properties. In patients with stroke, trunk control should be at a sufficient level in order to ensure functionality in the acute period. Muscle tone and viscoelasticity must be normal in order for trunk control to be at an adequate level. For this reason, in our study, the ability to control the trunk of patients with acute stroke will be associated with the viscoelastic properties of trunk muscles. Gaining a better understanding of changes in tissue distribution by looking at the viscoelasticity of trunk muscles and comparing them to the unaffected intact extremity will lead to better and more targeted interventions for rehabilitation.

The study will be carried out at Sanko University Sani Konukoğlu Practice and Research Hospital. Acute stroke patients who will voluntarily participate in the study will be included.

Inclusion criteria;

* Patients with ischemic cerebro-vascular disease within the first 72 hours,
* Patients with a National Institute of Health (NIH) score below 15
* No additional neurological and orthopedic problems
* Patients who do not have any inconvenience in sitting hemodynamically
* agree to participate in the study voluntarily Exclusion criteria;
* Patients who come to the service outside the first 72 hours
* Uncooperative patients
* patients who have had two or more strokes
* Those who have had a Trans Ischemic Attack (TIA)
* Refused to participate in the study Patients who are hospitalized from SANKO University Hospital Neurology Service will be included in the study. Socio-demographic information of the included patients will be obtained. Then, trunk impairment scale, which is a 17-item scale developed to evaluate trunk performance in stroke patients, will be used for trunk control . MyotonPro device will be used to measure the elasticity of Thoracis Longissimus, Lumbar Multifidus, Trapeze and Rectus Femoris muscles.

Demographic information form: this form is a form that evaluates the demographic information, contact information and general information of individuals.

Trunk impairment scale: It is a 17-parameter scale developed to evaluate trunk control in patients with neurological deficits . Existing sections in the scale; static sitting balance (GBÖ Static), dynamic sitting balance (GBÖ Dynamic) and coordination (GBÖ Coordination). The total score is a minimum of 0 and a maximum of 23 points and it is accepted that the higher score shows better performance. For the initial position in all items, the patients are asked to sit with the thighs parallel to the floor, feet in full contact with the ground, knees flexed to 90º, without back support, with the hands and forearms supported on the thighs. All items are repeated 3 times and the best performance of the patient is recorded. In between tests, the patient is given stimuli and verbal or visual feedback by the observer. A total score of 0 is given to individuals who cannot maintain the starting position for 10 seconds. A Turkish validity and reliability study of the GBS in stroke patients was performed .

MyotonPRO is a mobile, removable handheld myotonometer. This tool is noninvasive and provides a quantitative assessment of a muscle's viscoelastic properties. These properties are characterized by various parameters such as hardness, tone and elasticity. The probe of MyotonPRO delivers a short (15 ms), low intensity (0.58 N) mechanical impact/impact on the skin on the muscle. The response of the touch then generates a recorded signal and an internal software program generates an acceleration graph. Measurements of various viscoelastic muscle properties such as stiffness, tone, and elasticity are then extracted from this graph . Measurements of Thoracis Longissimus, Lumbar Multifidus, Trapeze and Rectus Femoris muscles will be recorded bilaterally, in 3-repetition measurements.

ELIGIBILITY:
Inclusion Criteria:

* Patients with ischemic cerebro-vascular disease within the first 72 hours,

  * Patients with a National Institute of Health (NIH) score below 15
  * No additional neurological and orthopedic problems
  * Patients who do not have any inconvenience in sitting hemodynamically
  * agree to participate in the study voluntarily

Exclusion Criteria:

* Patients who come to the service outside the first 72 hours
* Uncooperative patients
* patients who have had two or more strokes
* Those who have had a Trans Ischemic Attack (TIA)
* Refused to participate in the study

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2023-11-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
trunk disorder scale | 1 weeks
  It is a scale consisting of 17 parameters developed for the evaluation of trunk control in patients with neurological deficits (EK8). Existing sections in the scale; static sitting balance (GBÖ Static), dynamic sitting balance (GBÖ Dynamic) and coordination (GBÖ Coordination). The total score is a minimum of 0 and a maximum of 23 points and it is accepted that the higher score shows better performance. For the initial position in all items, the patients are asked to sit with the thighs parallel to the floor, feet in full contact with the ground, knees flexed to 90º, without back support, with the hands and forearms supported on the thighs. All items are repeated 3 times and the best performance of the patient is recorded. In between tests, the patient is given stimuli and verbal or visual feedback by the observer.
viscoelastic properties of muscle | 1 weeks
  MyotonPRO is a mobile, removable handheld myotonometer. This tool is noninvasive and provides a quantitative assessment of a muscle's viscoelastic properties. These properties are characterized by various parameters such as hardness, tone and elasticity. The probe of MyotonPRO delivers a short (15 ms), low intensity (0.58 N) mechanical impact/impact on the skin on the muscle. The response of the touch then generates a recorded signal and an internal software program generates an acceleration graph. Measurements of various viscoelastic muscle properties such as stiffness, tone and elasticity are then extracted from this graph. Measurements of Thoracis Longissimus, Lumbar Multifidus, Trapeze and Rectus Femoris muscles will be recorded bilaterally, in 3-repetition measurements.

CONTACTS AND LOCATIONS:
Locations (1):
- Sanko University, Gaziantep, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No